CLINICAL TRIAL: NCT01294813
Title: Bronchoscopy and Electric Impedance Tomography to Investigate the Influence of Bronchoscopy on Pulmonary Regional Ventilation Measurements by Electric Impedance Tomography (EIT)
Brief Title: Bronchoscopy and Electric Impedance Tomography (EIT) Pilot Study
Acronym: Broncho-EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Stefan Krueger, MD, Assistant Professor, PD Dr. med. Stefan Krueger, Medical Clinic 1, RWTH Aachen University Hospital, Section of Cardiology, Pneumology and Angiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Bronchoscopy- EIT
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Electric Impedance Tomography; Bronchoscopy; Change in Lung Impedance Due to Ventilation; Recruitment; Improvement the Treatment of the Patient
Keywords: Electric Impedance Tomography (EIT); Ventilation; Bronchoscopy; Lung Impedance; Recruitment
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoscopy-EIT (Experimental): Patients who routinely undergo bronchoscopy will be measured by EIT directly before, directly after and 10, 30, 60 minutes after bronchoscopy with a rubber belt which is placed around their chest. The EIT measurements will take 1-2 minutes; the total examination will last 1.5 hours.
  Interventions: Device: Electrical Impedance Tomography (EIT)

INTERVENTIONS:
Device: Electrical Impedance Tomography (EIT) — EIT measurements of 1-2 minutes are performed in patients who routinely undergo bronchoscopy (during 1.5 hours) before, directly after and 10, 30, 60 minutes after bronchoscopy. Therefore the rubber belt including 16 integrated electrographic electrodes is placed around the patient´s chest and connected with an EIT device. EIT data are generated by application of a small alternating current of 5mA and 50kHz and are stored and analyzed offline on a personal computer. Pseudonomyzed EIT data are evaluated descriptively.

SUMMARY:
Electrical Impedance Tomography (EIT)is a technique based on the injection of small currents and voltage measurements using electrodes on the skin surface generating cross-sectional images representing impedance change in a slice of the thorax. It is a radiation free, non-invasive and portable lung imaging technique. Impedance changes in lung ventilation are investigated in mechanically ventilated patients who routinely undergo bronchoscopy in intensive care medicine. Bronchoscopy is performed to suction secretions as well as to analyze the secretions to recognize inflammations and diseases. It is an essential intervention which causes changes in ventilation which remain for 1-2 hours. It is not completely investigated why these changes in ventilation remain for so long time and how they are distributed regionally. Therefore the purpose of this study is to investigate the change in pulmonary regional ventilation in patients who routinely undergo bronchoscopy to possibly generate ideas how to optimize the ventilation after bronchoscopy to optimize the patient´s treatment.

DETAILED DESCRIPTION:
In 20 mechanically ventilated patients who routinely undergo bronchoscopy Electrical Impedance Tomography (EIT) measurements whereby, evaluable data of 10 patients are needed, of about 1-2 minutes are performed directly before, directly after and 10, 30, and 60 minutes after bronchoscopy parallel to the following routine measurements: tidal volume, resistance, compliance, heart rate, blood pressure, SpO2 and blood gas values. Prior to the examination a rubber belt with 16 integrated electrocardiographic electrodes is placed around the thorax connected with an EIT- device. EIT data are generated by application of a small alternating current of 5mA and 50kHz and are stored and analyzed offline on a personal computer. The EIT provides a mapping of the distribution of the lung´s electrical impedance and exhibits a far temporal resolution of up to 40 tomograms per second. Because of electrical impedance of the pulmonal tissue is dependant to the air content, the air distribution within the lung over a certain period can be monitored. Analyzing the EIT- data it might be possible to explain the distribution in regional ventilation and how the ventilation could be optimized right after the bronchoscopy to optimize the patient´s treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients > 18 years old
* Mechanically ventilated patients who routinely undergo bronchoscopy

Exclusion Criteria:

* Pregnancy and Breastfeeding
* Active implants, heart pace makers and implanted converter defibrillator
* Foreign metallic objects in the thorax
* Cardiac valves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of the change in lung impedance due to ventilation before and after bronchoscopy by EIT measurements | Single Measurement of 1.5 hours
  It will be investigated if there are changes in lung impedance due to changes in ventilation before, directly after and 10, 30, 60 minutes after bronchoscopy in order to investigate their regional distribution and to generate ideas how the ventilation could be optimized to improve recruitment of the patient´s treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krueger, MD, Assoc. Prof., Principal Investigator — University Hospital Aachen, Medical Clinic 1, Section of Pneumology, 52074 Aachen, Nordrhein-Westfalen, Germany
Locations (1):
- Faculty Medical Clinic 1, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany